CLINICAL TRIAL: NCT07338175
Title: Efficacy and Safety of Minocycline in Patients With Acute Spontaneous Intracerebral Hemorrhage: A Prospective, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group, Phase III Trial
Brief Title: Efficacy and Safety of Minocycline in Acute Spontaneous Intracerebral Hemorrhage
Acronym: MISTICH
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Xingquan Zhao, Xingquan Zhao; Yilong Wang, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MISTICH
Record Dates: First submitted 2026-01-03; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Intracerebral Hemorrhage
Keywords: Intracerebral Hemorrhage; Minocycline; Neuroprotection
MeSH Terms: conditions — Cerebral Hemorrhage; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Comparator: Minocycline treatment group (Experimental): Minocycline Hydrochloride Capsules (50 mg per capsule). The first dose (200mg, 4 capsules) should be given immediately after randomization (within 30 minutes); Subsequently, 100mg (2 capsules) will be administered once every 12 hours; a total of 10 times (lasting 5 days; the subject with dysphagia will be administrated through a nasal feeding tube).
  Interventions: Drug: Minocycline hydrochloride capsules
- Placebo Comparator: Minocycline placebo-control group (Placebo Comparator): Placebo of Minocycline Hydrochloride capsules (50mg per capsule, containing 0 mg of Minocycline). The method of administration was the same as that of treatment group.
  Interventions: Drug: Placebo capsules of Minocycline hydrochloride capsules

INTERVENTIONS:
Drug: Minocycline hydrochloride capsules — 50 mg per capsule, containing 50mg of Minocycline Hydrochloride
  Arms: Active Comparator: Minocycline treatment group
Drug: Placebo capsules of Minocycline hydrochloride capsules — 50 mg per capsule, containing 0 mg of Minocycline Hydrochloride
  Arms: Placebo Comparator: Minocycline placebo-control group

SUMMARY:
This is a prospective, multicenter, randomized, double-blind, placebo-controlled clinical trial. It aims to evaluate the efficacy and safety of oral minocycline in patients with acute spontaneous intracerebral hemorrhage within 48 hours of onset.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the efficacy and safety of 5-day Minocycline versus placebo in patients with acute intracerebral hemorrhage within 48 hours of onset. In addition, we will explore the effect of Minocycline versus placebo on indicators of venous neuroinflammation at different time points in patients with acute intracerebral hemorrhage within 48 hours of onset.

A total of 1192 participants will be randomized 1:1 to receive either minocycline or matching placebo for 5 days, in addition to guideline-based standard medical care.

The primary objective is to evaluate the effect of Minocycline in improving the level of 90-day mRS score to 0-3 in patients with acute intracerebral hemorrhage within 48 hours of onset.

The trial is divided into three phases: screening/baseline period, treatment period, and follow-up period. The visit schedule is as follows: Randomized participants are interviewed at screening/baseline period, 72±12 hours, 7±1 days, 90±7 days,180±7 days after randomization, and when events occur.

ELIGIBILITY:
Inclusion Criteria:

1. CT-confirmed spontaneous supratentorial intracerebral hemorrhage;
2. Aged 18 to 80 years;
3. Within 48 hours of symptom onset;
4. Hematoma volume 15-40 ml;
5. NIHSS score 8-24, with item 1a ≤ 2;
6. Signed informed consent by the patient or legal representative.

Exclusion Criteria:

1. Secondary intracerebral hemorrhage (traumatic, tumor-related, vascular malformation, aneurysm, coagulation disorder, etc.);
2. Intraventricular hemorrhage filling one entire lateral ventricle, third ventricle, or fourth ventricle, or more than half of two lateral ventricles;
3. Significant subarachnoid hemorrhage (Fisher grade ≥ 3) or subdural hemorrhage;
4. Patients with uncontrollable hypertension or those at high risk of hematoma expansion indicated by imaging signs;
5. Progressive neurological or other severe systemic diseases;
6. Planned surgical intervention for the intracerebral hemorrhage;
7. Pre-stroke disability (modified Rankin Scale score > 1);
8. Severe cardiac insufficiency (NYHA Class III-IV), severe liver disease (ALT or AST > 3 times the normal upper limit value), severe renal insufficiency (serum creatinine > 2 times the normal upper limit value, or glomerular filtration rate < 45 ml/min), or malignancy with life expectancy < 1 year;
9. Moderate to severe anemia (hemoglobin < 90 g/L), thrombocytopenia (platelet count < 100×10^9/L), leukopenia (white blood cell count < 2×10^9/L), or coagulopathy (INR > 1.5);
10. Allergy or intolerance to minocycline or other tetracycline antibiotics;
11. History of pseudomembranous enteritis or antibiotic-associated enteritis;
12. Use of tetracycline antibiotics within the past week;
13. Intracranial or spinal surgery within the past 3 months;
14. Any major surgery or severe physical trauma within the past month;
15. Females who are pregnant, within 30 days postpartum, or in the lactation period.
16. Participated in other interventional clinical trials within the past 3 months;
17. Inability to obtain signed informed consent from the patient or representative;
18. Other conditions that are not suitable for participating in this clinical trial, such as inability to understand and/or follow the research procedures due to mental, cognitive, emotional, or physical disorders, etc.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1192 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
mRS score 0-3 | At 90±7 days after randomization
  Modified Rankin Scale score

SECONDARY OUTCOMES:
mRS score | At 90±7 days and 180±7 days after randomization
  Modified Rankin Scale score
Changes in NIHSS score compared with baseline score | At 72±12 hours and 7±1 days after randomization
  NIHSS score
Changes in Glasgow Coma Scale score compared with baseline score | At 72±12 hours and 7±1 days after randomization
  Glasgow Coma Scale score
Early neurological deterioration | At 72±12 hours and 7±1 days after randomization
  Early neurological deterioration is defined as a decrease of ≥2 in GCS score or an increase of ≥4 in NIHSS score caused by non-sedatives/sleeping drugs compared with the baseline level.
Changes in hs-CRP level compared with baseline level | At 72±12 hours and 7±1 days after randomization
  hs-CRP is examined to evaluate the level of systematic inflammation.
Volume of perihematomal edema (PHE) | At 7±1 days after randomization
  Volume of perihematomal edema (PHE) on MRI
EQ-5D-5L utility score | At 90±7 days and 180±7 days after randomization
  Quality of life assessed by the EQ-5D-5L utility score
Recurrent stroke | At 90±7 days and 180±7 days after randomization
  Recurrent stroke includes ischemic stroke and hemorrhagic stroke.
Combined vascular events | At 90±7 days and 180±7 days after randomization
  Combined vascular events include stroke, myocardial infarction, and vascular death.

OTHER OUTCOMES:
Changes in the levels of venous neuroinflammation indicators compared with baseline levels | At 72±12 hours and 7±1 days after randomization
  Venous neuroinflammation indicators (IL, TNF-α, TGF-β, NFL, etc.)
Perihematomal blood-brain barrier permeability | At 7±1 days after randomization
  Perihematomal blood-brain barrier permeability is assessed using dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI).
Hematoma expansion or rebleeding | At 72±12 hours and 7±1 days after randomization
  Hematoma expansion or rebleeding
Antibiotic-associated diarrhea, enteritis, and constipation | At 7±1 days after randomization
  Antibiotic-associated diarrhea, enteritis, and constipation
Any bleeding events | At 90±7 days after randomization
  Any bleeding events
Adverse events (AE) | At 90±7 days after randomization
  Adverse events (AE)
Serious adverse events (SAE) | At 90±7 days after randomization
  Serious adverse events (SAE)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Chang JJ, Kim-Tenser M, Emanuel BA, Jones GM, Chapple K, Alikhani A, Sanossian N, Mack WJ, Tsivgoulis G, Alexandrov AV, Pourmotabbed T. Minocycline and matrix metalloproteinase inhibition in acute intracerebral hemorrhage: a pilot study. Eur J Neurol. 2017 Nov;24(11):1384-1391. doi: 10.1111/ene.13403. Epub 2017 Sep 20. PMID 28929560
- [Result] Lu Y, Guan L, Zhang M, Yang Q, Qiu B, Zhou D, Wang Y, Pan Y, Wang L, Zhou X, Qu H, Liao X, Liu L, Zhao X, Bath PM, Johnston SC, Amarenco P, Wang Y, Wang Y. Rationale and Study Design to Assess the Efficacy and Safety of Minocycline in Patients with Moderate to Severe Acute Ischaemic Stroke (EMPHASIS). Stroke Vasc Neurol. 2025 Dec 23;10(6):786-792. doi: 10.1136/svn-2024-003577. PMID 40147820
- [Result] Fouda AY, Newsome AS, Spellicy S, Waller JL, Zhi W, Hess DC, Ergul A, Edwards DJ, Fagan SC, Switzer JA. Minocycline in Acute Cerebral Hemorrhage: An Early Phase Randomized Trial. Stroke. 2017 Oct;48(10):2885-2887. doi: 10.1161/STROKEAHA.117.018658. Epub 2017 Sep 8. PMID 28887388
- [Result] Lampl Y, Boaz M, Gilad R, Lorberboym M, Dabby R, Rapoport A, Anca-Hershkowitz M, Sadeh M. Minocycline treatment in acute stroke: an open-label, evaluator-blinded study. Neurology. 2007 Oct 2;69(14):1404-10. doi: 10.1212/01.wnl.0000277487.04281.db. PMID 17909152
- [Result] Wu DC, Jackson-Lewis V, Vila M, Tieu K, Teismann P, Vadseth C, Choi DK, Ischiropoulos H, Przedborski S. Blockade of microglial activation is neuroprotective in the 1-methyl-4-phenyl-1,2,3,6-tetrahydropyridine mouse model of Parkinson disease. J Neurosci. 2002 Mar 1;22(5):1763-71. doi: 10.1523/JNEUROSCI.22-05-01763.2002. PMID 11880505
- [Result] Kraus RL, Pasieczny R, Lariosa-Willingham K, Turner MS, Jiang A, Trauger JW. Antioxidant properties of minocycline: neuroprotection in an oxidative stress assay and direct radical-scavenging activity. J Neurochem. 2005 Aug;94(3):819-27. doi: 10.1111/j.1471-4159.2005.03219.x. PMID 16033424
- [Result] Lee JM, Yin K, Hsin I, Chen S, Fryer JD, Holtzman DM, Hsu CY, Xu J. Matrix metalloproteinase-9 in cerebral-amyloid-angiopathy-related hemorrhage. J Neurol Sci. 2005 Mar 15;229-230:249-54. doi: 10.1016/j.jns.2004.11.041. Epub 2004 Dec 29. PMID 15760647
- [Result] Yrjanheikki J, Tikka T, Keinanen R, Goldsteins G, Chan PH, Koistinaho J. A tetracycline derivative, minocycline, reduces inflammation and protects against focal cerebral ischemia with a wide therapeutic window. Proc Natl Acad Sci U S A. 1999 Nov 9;96(23):13496-500. doi: 10.1073/pnas.96.23.13496. PMID 10557349
- [Result] Garrido-Mesa N, Zarzuelo A, Galvez J. What is behind the non-antibiotic properties of minocycline? Pharmacol Res. 2013 Jan;67(1):18-30. doi: 10.1016/j.phrs.2012.10.006. Epub 2012 Oct 17. PMID 23085382
- [Result] Fu Y, Hao J, Zhang N, Ren L, Sun N, Li YJ, Yan Y, Huang D, Yu C, Shi FD. Fingolimod for the treatment of intracerebral hemorrhage: a 2-arm proof-of-concept study. JAMA Neurol. 2014 Sep;71(9):1092-101. doi: 10.1001/jamaneurol.2014.1065. PMID 25003359
- [Result] Xue M, Yong VW. Neuroinflammation in intracerebral haemorrhage: immunotherapies with potential for translation. Lancet Neurol. 2020 Dec;19(12):1023-1032. doi: 10.1016/S1474-4422(20)30364-1. PMID 33212054
- [Result] Bai Q, Xue M, Yong VW. Microglia and macrophage phenotypes in intracerebral haemorrhage injury: therapeutic opportunities. Brain. 2020 May 1;143(5):1297-1314. doi: 10.1093/brain/awz393. PMID 31919518
- [Result] Puy L, Perbet R, Figeac M, Duchene B, Deramecourt V, Cordonnier C, Berezowski V. Brain Peri-Hematomal Area, a Strategic Interface for Blood Clearance: A Human Neuropathological and Transcriptomic Study. Stroke. 2022 Jun;53(6):2026-2035. doi: 10.1161/STROKEAHA.121.037751. Epub 2022 Apr 25. PMID 35465695
- [Result] Li N, Guo J, Kang K, Zhang J, Zhang Z, Liu L, Liu X, Du Y, Wang Y, Zhao X. Cytotoxic Edema and Adverse Clinical Outcomes in Patients with Intracerebral Hemorrhage. Neurocrit Care. 2023 Apr;38(2):414-421. doi: 10.1007/s12028-022-01603-2. Epub 2022 Sep 30. PMID 36180765
- [Result] Cordonnier C, Demchuk A, Ziai W, Anderson CS. Intracerebral haemorrhage: current approaches to acute management. Lancet. 2018 Oct 6;392(10154):1257-1268. doi: 10.1016/S0140-6736(18)31878-6. PMID 30319113
- [Result] Greenberg SM, Ziai WC, Cordonnier C, Dowlatshahi D, Francis B, Goldstein JN, Hemphill JC 3rd, Johnson R, Keigher KM, Mack WJ, Mocco J, Newton EJ, Ruff IM, Sansing LH, Schulman S, Selim MH, Sheth KN, Sprigg N, Sunnerhagen KS; American Heart Association/American Stroke Association. 2022 Guideline for the Management of Patients With Spontaneous Intracerebral Hemorrhage: A Guideline From the American Heart Association/American Stroke Association. Stroke. 2022 Jul;53(7):e282-e361. doi: 10.1161/STR.0000000000000407. Epub 2022 May 17. No abstract available. PMID 35579034
- [Result] Wu TY, Sharma G, Strbian D, Putaala J, Desmond PM, Tatlisumak T, Davis SM, Meretoja A. Natural History of Perihematomal Edema and Impact on Outcome After Intracerebral Hemorrhage. Stroke. 2017 Apr;48(4):873-879. doi: 10.1161/STROKEAHA.116.014416. Epub 2017 Mar 8. PMID 28275199
- [Result] Murthy SB, Moradiya Y, Dawson J, Lees KR, Hanley DF, Ziai WC; VISTA-ICH Collaborators. Perihematomal Edema and Functional Outcomes in Intracerebral Hemorrhage: Influence of Hematoma Volume and Location. Stroke. 2015 Nov;46(11):3088-92. doi: 10.1161/STROKEAHA.115.010054. Epub 2015 Sep 22. PMID 26396030
- [Result] Sheth KN. Spontaneous Intracerebral Hemorrhage. N Engl J Med. 2022 Oct 27;387(17):1589-1596. doi: 10.1056/NEJMra2201449. No abstract available. PMID 36300975
- [Result] Gross BA, Jankowitz BT, Friedlander RM. Cerebral Intraparenchymal Hemorrhage: A Review. JAMA. 2019 Apr 2;321(13):1295-1303. doi: 10.1001/jama.2019.2413. PMID 30938800
- [Result] Wang WJ, Lu JJ, Wang YJ, Wang CX, Wang YL, Hoff K, Yang ZH, Liu LP, Wang AX, Zhao XQ; China National Stroke Registry (CNSR). Clinical characteristics, management, and functional outcomes in Chinese patients within the first year after intracerebral hemorrhage: analysis from China National Stroke Registry. CNS Neurosci Ther. 2012 Sep;18(9):773-80. doi: 10.1111/j.1755-5949.2012.00367.x. PMID 22943144
- [Result] Flower O, Smith M. The acute management of intracerebral hemorrhage. Curr Opin Crit Care. 2011 Apr;17(2):106-14. doi: 10.1097/MCC.0b013e328342f823. PMID 21169826
- [Result] Zhao Y, Hua X, Ren X, Ouyang M, Chen C, Li Y, Yin X, Song P, Chen X, Wu S, Song L, Anderson CS. Increasing burden of stroke in China: A systematic review and meta-analysis of prevalence, incidence, mortality, and case fatality. Int J Stroke. 2023 Mar;18(3):259-267. doi: 10.1177/17474930221135983. Epub 2022 Nov 16. PMID 36274585
- [Result] Ma Q, Li R, Wang L, Yin P, Wang Y, Yan C, Ren Y, Qian Z, Vaughn MG, McMillin SE, Hay SI, Naghavi M, Cai M, Wang C, Zhang Z, Zhou M, Lin H, Yang Y. Temporal trend and attributable risk factors of stroke burden in China, 1990-2019: an analysis for the Global Burden of Disease Study 2019. Lancet Public Health. 2021 Dec;6(12):e897-e906. doi: 10.1016/S2468-2667(21)00228-0. PMID 34838196
- [Result] GBD 2019 Stroke Collaborators. Global, regional, and national burden of stroke and its risk factors, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet Neurol. 2021 Oct;20(10):795-820. doi: 10.1016/S1474-4422(21)00252-0. Epub 2021 Sep 3. PMID 34487721